CLINICAL TRIAL: NCT01214525
Title: The Improvement in Uroflow and Postvoid Residual Urine After Urethral Meatotomy in Children With Meatal Stenosis
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10144-2010CTIL
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Urethral Meatal Stenosis
Keywords: Meatal stenosis; Meatotomy; Uroflow; Postvoid residual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Meatotomy: Toilet trained children scheduled for urethral meatotomy for the treatment of urethral meatal stenosis.

SUMMARY:
The improvement in uroflow and postvoid residual urine in children after urethral meatotomy for meatal stenosis. The hypothesis is that there is an improvement in both parameters, thus justifying the procedure.

DETAILED DESCRIPTION:
Urethral meatal stenosis is a known complication of circumcision occuring in up to 3% of newborns undergoing circumcision. It is customary to perform a meatotomy in order to prevent bladder outlet obstruction, although bladder outlet obstruction has never been proven and improvement has only been proved in a single, small, retrospective study. Our intention is to evaluate the improvement in objective parameters (uroflow and postvoid residual urine) after urethral meatotomy by measuring these parameter before the procedure, one month after the procedure and one year after the procedure. Symptoms assessment will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Toilet trained children
* Before puberty
* No other urologic disease that might affect the measurements
* Primary (first) repair

Exclusion Criteria:

* Children unable to urinate on command
* Children that have started their sexual puberty
* Children with other urologic disease that might affect the study measurements
* Recurrent stenosis after previous repair

Ages: 2 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Toilet trained children, before puberty, scheduled for urethral meatotomy for the treatment of urethral meatal stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08-01 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
Improved maximal urine flow | one month and one year

SECONDARY OUTCOMES:
Improved (reduced) postvoid residual urine | One month and one year

CONTACTS AND LOCATIONS:
Overall Officials: Itay A Sternberg, MD, Principal Investigator — Meir Medical Center; Amos Neheman, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] VanderBrink BA, Gitlin J, Palmer LS. Uroflowmetry parameters before and after meatoplasty for primary symptomatic meatal stenosis in children. J Urol. 2008 Jun;179(6):2403-6; discussion 2406. doi: 10.1016/j.juro.2008.01.169. Epub 2008 Apr 23. PMID 18436251